CLINICAL TRIAL: NCT06176508
Title: A Randomized, Double-blind, Placebo- and Comparator-controlled, Multicenter, Phase 2 Trial to Assess the Efficacy and Safety of HS-10374 in Adults With Active Psoriatic Arthritis
Brief Title: Efficacy and Safety of HS-10374 Compared to Placebo in Adults With Active Psoriatic Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10374-202
Record Dates: First submitted 2023-12-08; First posted 2023-12-19 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-10374 Dose 1 (Experimental)
  Interventions: Drug: HS-10374
- HS-10374 Dose 2 (Experimental)
  Interventions: Drug: HS-10374
- Placebo (Placebo Comparator)
  Interventions: Drug: HS-10374-matched placebo tablets
- tofacitinib (Active Comparator)
  Interventions: Drug: Tofacitinib 5Mg Tab,Oral

INTERVENTIONS:
Drug: HS-10374 — Administered orally QD for 16 weeks
  Arms: HS-10374 Dose 1; HS-10374 Dose 2
Drug: HS-10374-matched placebo tablets — Administered orally QD for 16 weeks
  Arms: Placebo
Drug: Tofacitinib 5Mg Tab,Oral — Administered orally BID for 16 weeks
  Arms: tofacitinib

SUMMARY:
This study has been designed to explore the clinical efficacy and safety of HS-10374 in the treatment of active psoriatic arthritis. Additionally, this study is to find the optimal dosing for the future clinical development of HS-10374.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18-75 years.
2. Has a history of psoriatic arthritis (PsA) for at least 6 months, and meets the Classification Criteria for Psoriatic Arthritis (CASPAR) at screening.
3. Active arthritis as shown ≥ 3 swollen joints (66 joints) and ≥ 3 tender joints (68 joints) at both screening and baseline.
4. Active plague psoriatic skin lesion or documented history of plague psoriatic at screening.
5. hs-CRP ≥ 3mg/L at screening.
6. Subjects either (i) do not have prior exposure to biologics (biologic-naïve) or (ii) have failed or been intolerant to 1 TNF-inhibitor (TNFi-experienced).

Exclusion Criteria:

1. Non-plaque psoriasis (ie, guttate, inverse, pustular, erythrodermic or drug-induced psoriasis), with the exception of nail psoriasis, which is allowed.
2. Other autoimmune or autoinflammatory condition ( ie, rheumatoid arthritis, systemic lupus erythematous, gout), with the exception of inflammatory bowel disease and/or autoimmune uveitis being inactive at least 12 months before the screening, as assessed by the investigator.
3. Active fibromyalgia syndrome
4. Recent history of active infection, chronic infection history or risk of serious infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants meeting American College of Rheumatology improvement of 20% (ACR20) response at Week 16 | At week 16
  The ACR 20, ACR 50 or ACR 70 definition of improvement is a 20%, 50% or 70% improvement, respectively, over baseline in tender and swollen joint counts and a 20%, 50% or 70% improvement, respectively, in 3 of the 5 remaining core data set measures (Subject Global Assessment of disease activity, Physician Global Assessment of psoriatic arthritis, Subject global assessment of pain, HAQ-DI, hs-CRP).

SECONDARY OUTCOMES:
Proportion of participants meeting American College of Rheumatology improvement of 20% (ACR20) response at Week 12 | At week 12
  The ACR 20, ACR 50 or ACR 70 definition of improvement is a 20%, 50% or 70% improvement, respectively, over baseline in tender and swollen joint counts and a 20%, 50% or 70% improvement, respectively, in 3 of the 5 remaining core data set measures (Subject Global Assessment of disease activity, Physician Global Assessment of psoriatic arthritis, Subject global assessment of pain, HAQ-DI, hs-CRP).
Proportion of participants meeting American College of Rheumatology improvement of 50% (ACR50) response at Week 16 | At week 16
  The ACR 20, ACR 50 or ACR 70 definition of improvement is a 20%, 50% or 70% improvement, respectively, over baseline in tender and swollen joint counts and a 20%, 50% or 70% improvement, respectively, in 3 of the 5 remaining core data set measures (Subject Global Assessment of disease activity, Physician Global Assessment of psoriatic arthritis, Subject global assessment of pain, HAQ-DI, hs-CRP).
Proportion of participants meeting American College of Rheumatology improvement of 70% (ACR70) response at Week 16 | At week 16
  The ACR 20, ACR 50 or ACR 70 definition of improvement is a 20%, 50% or 70% improvement, respectively, over baseline in tender and swollen joint counts and a 20%, 50% or 70% improvement, respectively, in 3 of the 5 remaining core data set measures (Subject Global Assessment of disease activity, Physician Global Assessment of psoriatic arthritis, Subject global assessment of pain, HAQ-DI, hs-CRP).
Change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) score at week 16 | At week 16
  The HAQ-DI is a patient-reported outcome measure that assesses the degree of difficulty a subject has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. For reach item in the questionnaire the level of activity is cored from 0 to 3 with 0 representing "no difficulty", 1 as "some difficulty", 2 as much "difficulty", and 3 has "unable to do". Any activity that requires assistance from another individual or requires the use of an assistive device adjusts to a score of 2 or more.
Proportion of participants meeting Psoriasis Area and Severity Index (PASI) 75/90 responses at week 16 | At week 16
  Psoriasis Area and Severity Index (PASI) is a scoring system quantifying the severity of psoriasis based on both lesion severity and area of involvement. PASI assessment is performed by investigators, and the numeric score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75, PASI 90 responses are defined as 75% or 90% improvement in PASI score from baseline.
Proportion of participants meeting Static physician's global assessment (sPGA) 0/1 score at week 16 | At week 16
  Static physician's global assessment (sPGA) of psoriasis is an average assessment of all psoriatic lesions based on erythema, induration, and scale. It's a 5-point scale performed by investigators. A sPGA score of 0 or 1 means "clear" or "almost clear" respectively.
Change from baseline in Psoriasis body surface area (BSA) at week 16 | At week 16
  Psoriasis body surface area (BSA) involvement is measured using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved.
Change from baseline in the dermatology life quality index (DLQI) scores at week 16 | At week 16
  The dermatology life quality index (DLQI) is a patient reported outcome measurement. It's a questionnaire consisting of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. Each question is scored on a scale of 0 to 3, and the sum of each scores range from 0 (no impairment of life quality) to 30 (maximum impairment).
Change from baseline in Disease Activity Score 28 with C-reactive protein (DAS28-CRP) score at week 16 | At week 16
  DAS28-CRP is a composite outcome measure that assesses: Numbers of joints in the hands (including metacarpophalangeal and proximal interphalangeal joints, except for distal interphalangeal joints), wrists, elbows, shoulders, and knees are swollen and/or tender over a total of 28; Hypersensitive-CRP in the blood to measure the degree of inflammation; Subject Global Assessment of disease activity.
  The results are combined to produce the DAS28-CRP score, which correlates with the extent of disease activity: ≤2.6: Disease remission; 2.6 - 3.2: Low disease activity; 3.2 - 5.1: Moderate disease activity; >5.1: High disease activity.
Change from baseline in the Disease Activity Index for Psoriatic Arthritis Score (DAPSA) at week 16 | At week 16
  The Disease Activity Index for Psoriatic Arthritis Score (DAPSA) is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender/painful joint count, swollen joint count, Subject Global Assessment of disease activity, Subject Global Assessment of pain, and hs-CRP.
Proportion of participants meeting Minimal Disease Activity (MDA) response at week 16 | At week 16
  Minimal Disease Activity (MDA) response is defined as a subject fulfilling 5 of 7 of the following outcomes: tender joint count ≤ 1; swollen joint count ≤ 1; PASI ≤ 1 or body surface area (BSA) ≤ 3%; Subject Global Assessment of pain ≤ 15; Subject Global Assessment of disease activity ≤ 20; HAQ-DI ≤ 0.5; Tender entheseal points ≤ 1
Change from baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) at week 16 | At week 16
  A composite measure calculated from the Physician Global Assessment of psoriatic arthritis, the Subject Global Assessment of disease activity, the Short Form Health Survey-36 Item (SF-36) Physical Component Summary (PCS), the swollen joint count, the tender joint count, the LEI, the tendor dactylitis count and the hs-CRP.
Proportion of participants achieving Psoriatic Arthritis Response Criteria (PsARC) at week 16 | At week 16
  The Psoriatic Arthritis Response Criteria (PsARC) consists of 4 measurements: tender/painful joint count, swollen joint count, Physician Global Assessment of psoriatic arthritis, and Subject Global Assessment of psoriatic arthritis. In order to be classified as a PsARC responder, subjects must achieve improvement in 2 of 4 measures, one of which must be joint pain or swelling, without worsening in any measure.
Change from baseline in the Short Form-36 Survey (SF-36) score at week 16 | At week 16
  The SF-36 is a patient-reported outcome measure in clinical practice and research. The instrument includes 36 items to measure the following 8 health dimensions over the past 4 week: 1) limitations in physical activities, such as bathing or dressing; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality; and 8) general health perceptions.
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score among participants with spondylitis as one of their presentations of PsA at week 16 | At week 16
  Symptoms of spondylitis over the past week will be evaluated using the BASDAI, which consists of a 0 to 100 scale measuring discomfort, pain, and fatigue in response to 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis:
  * Fatigue
  * Spinal pain
  * Joint pain and swelling
  * Areas of localized tenderness
  * Morning stiffness duration
  * Morning stiffness severity A higher count indicates worse disease.
Change from baseline in dactylitis by Leed's dactylitis index (LDI) at week 16 | At week 16
  Leed's Dactylitis Index (LDI) is a quantitative measurement of dactylitis in the 20 digits using a dactylometer. The circumference of the affected and contralateral digits, and tenderness of the affected digits are measured to generate a total score. A higher score indicates worse dactylitis and is based on the current evaluation.
Change from baseline in enthesitis by Leed's enthesitis index (LEI) at week 16 | At week 16
  The Leed's enthesitis index (LEI) was developed specifically for PsA. An overall score of 0 to 6 is derived from the presence or absence of tenderness at 6 entheseal sites (right and left: lateral epicondyle, medial femoral condyle, and Achilles tendon insertion) at the time of evaluation. A higher count indicates a greater enthesitis burden.
Incidence of adverse events (AEs), serious adverse events (SAEs) | Baseline to Week 20
Ctrough of HS-10374 | Baseline to Week 16
  Trough observed plasma concentration of HS-10374

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China